CLINICAL TRIAL: NCT00529529
Title: A 26-week Treatment, Randomized, Multicenter, Double-blind, Double-dummy, Parallel-group Study to Assess the Safety of Indacaterol (300 and 600 µg o.d.) in Patients With Moderate to Severe Persistent Asthma, Using Salmeterol (50 µg b.i.d.) as an Active Control
Brief Title: Safety of Indacaterol in Patients (≥ 12 Years) With Moderate to Severe Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2338
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2011-08-19 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Asthma
Keywords: asthma; QAB149; indacaterol
MeSH Terms: conditions — Asthma | interventions — indacaterol; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Indacaterol 300 μg (Experimental): Patients received indacaterol 300 μg delivered via a single dose dry powder inhaler (SDDPI) once daily (od) in the morning (between 07:00 and 11:00 AM). In addition to indacaterol 300 μg, patients received indacaterol and salmeterol placebo inhalations in the morning and salmeterol placebo inhalation in the evening (between 7:00 and 11:00 PM). Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 300 μg; Drug: Placebo to indacaterol; Drug: Placebo to salmeterol
- Indacaterol 600 μg (Experimental): Patients received indacaterol 600 μg (2 x 300 μg capsules) delivered via single dose dry powder inhalers (SDDPI) once daily (od) in the morning (between 07:00 and 11:00 AM). In addition to indacaterol 600 μg, patients received salmeterol placebo inhalation in the morning and the evening (between 7:00 and 11:00 PM). Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 300 μg; Drug: Placebo to salmeterol
- Salmeterol 50 μg (Active Comparator): Patients received salmeterol 50 μg delivered via the salmeterol proprietary dry powder inhalation device bis in die (bid, twice daily), once in the morning (between 07:00 and 11:00 AM) and once in the evening (between 7:00 and 11:00 PM). In addition to salmeterol 50 μg, patients received 2 indacaterol placebo inhalations in the morning. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Salmeterol 50 μg; Drug: Placebo to indacaterol

INTERVENTIONS:
Drug: Indacaterol 300 μg — Indacaterol was supplied as powder filled capsules together with a single dose dry powder inhaler (SDDPI).
  Arms: Indacaterol 300 μg; Indacaterol 600 μg
Drug: Salmeterol 50 μg — Salmeterol was supplied as powder filled capsules together with the manufacturer's proprietary dry powder inhalation device.
  Arms: Salmeterol 50 μg
Drug: Placebo to indacaterol — Placebo to indacaterol was supplied as powder filled capsules together with a single dose dry powder inhaler (SDDPI).
  Arms: Indacaterol 300 μg; Salmeterol 50 μg
Drug: Placebo to salmeterol — Placebo to salmeterol was supplied as powder filled capsules together with the manufacturer's proprietary dry powder inhalation device.
  Arms: Indacaterol 300 μg; Indacaterol 600 μg

SUMMARY:
This study was designed to assess the safety of indacaterol (300 µg and 600 µg (2 x 300 μg capsules) once daily [od]), compared with salmeterol (50 μg twice a day [b.i.d.]), over 26 weeks, in patients with moderate to severe persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥ 12 years (or ≥ 18 years depending upon regulatory and/or Institutional Review Board/Independent Ethics Committee/Research Ethics Board [IRB/IEC/REB] approval) who have signed an informed consent form.
2. Patients with moderate to severe persistent asthma, diagnosed according to the Global Initiative for Asthma (GINA) guidelines (Updated 2006) and who additionally meet the following criteria:

   * Patients who have used treatment with a bronchodilator, either regularly or on-demand, and who had used a daily dose of at least 100 μg beclomethasone dipropionate (or equivalent) for at least 1 month prior to screening.
   * Patients whose forced expiratory volume in 1 second (FEV1) is ≥ 50% of the predicted normal value.
   * Patients with documented (in the previous 6 months) or who demonstrate (prior to randomization) a ≥ 12% and at least 200 ml increase in FEV1, after inhaling 200 μg salbutamol.

Exclusion Criteria:

1. Pregnant or nursing (lactating) women and women of child-bearing potential UNLESS they meet pre-specified definitions of post-menopausal or are using pre-specified acceptable methods of contraception.
2. Patients who have used tobacco products within the 12 month period prior to screening, or who have a smoking history of greater than 10 pack years.
3. Patients who suffer from chronic obstructive pulmonary disease (COPD) as diagnosed by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines (2006).
4. Patients who have had emergency room treatment for an acute asthma attack in the 6 weeks prior to screening or who have been hospitalized for an acute asthma attack in the 6 months prior to screening, or at any time between screening and Week 1.
5. Patients with diabetes Type I or those with uncontrolled diabetes Type II including patients with a history of blood glucose levels consistently outside the normal range or glycosylated hemoglobin (HbA1C) > 8.0% measured at screening.
6. Patients who, in the judgment of the investigator or the responsible Novartis personnel, have a clinically significant condition or a clinically relevant laboratory abnormality that might compromise patient safety or compliance, interfere with evaluation, or preclude completion of the study.
7. Patients with a history of long QT syndrome, or whose QTc interval (Bazett's formula) is prolonged to > 450 ms (males) or > 470 ms (females).
8. Certain medications for asthma and allied conditions such as long-acting bronchodilators must not be used prior to screening and for a pre-specified minimum washout period.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 805 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (119):
- United States (49):
  - Novartis Investigator Site, Glendale, Arizona
  - Novartis Investigator Site, Phoenix, Arizona
  - Novartis Investigator Site, Encinitas, California
  - Novartis Investigator Site, Huntington Beach, California
  - Novartis Investigator Site, Long Beach, California
  - Novartis Investigator Site, Los Angeles, California
  - Novartis Investigator Site x 2 sites, Oakland, California
  - Novartis Investigator Site, Orange, California
  - Novartis Investigator Site, Palmdale, California
  - Novartis Investigator Site, San Diego, California
  - Novartis Investigator Site, Walnut Creek, California
  - Novartis Investigator Site, Denver, Colorado
  - Novartis Investigator Site, Englewood, Colorado
  - Novartis Investigator Site, Lakewood, Colorado
  - Novartis Investigator Site, Brandon, Florida
  - Novartis Investigator Site, Largo, Florida
  - Novartis Investigator Site, Miami, Florida
  - Novartis Investigator Site, Panama City, Florida
  - Novartis Investigator Site, Pensacola, Florida
  - Novartis Investigator Site x 2 sites, Pensacola, Florida
  - Novartis Investigator Site, Tamarac, Florida
  - Novartis Investigator Site, Albany, Georgia
  - Novartis Investigator Site, Stockbridge, Georgia
  - Novartis Investigator Site, Overland Park, Kansas
  - Novartis Investigator Site, Topeka, Kansas
  - Novartis Investigator Site, Florence, Kentucky
  - Novartis Investigator Site, Baltimore, Maryland
  - Novartis Investigator Site, Wheaton, Maryland
  - Novartis Investigator Site, North Dartmouth, Massachusetts
  - Novartis Investigator Site, Ann Arbor, Michigan
  - Novartis Investigator Site, Ypsilanti, Michigan
  - Novartis Investigator Site, Springfield, Missouri
  - Novartis Investigator Site, St Louis, Missouri
  - Novartis Investigator Site, Omaha, Nebraska
  - Novartis Investigator Site, Northfield, New Jersey
  - Novartis Investigator Site, Rockville Centre, New York
  - Novartis Investigator Site, Charlotte, North Carolina
  - Novartis Investigator Site, High Point, North Carolina
  - Novartis Investigator Site, Winston-Salem, North Carolina
  - Novartis Investigator Site, Cincinnati, Ohio
  - Novartis Investigator Site, Toledo, Ohio
  - Novartis Investigator Site, Edmond, Oklahoma
  - Novartis Investigator Site, Oklahoma City, Oklahoma
  - Novartis Investigator Site, Greenville, South Carolina
  - Novartis Investigator Site, Dallas, Texas
  - Novartis Investigator site, Houston, Texas
  - Novartis Investigator Site, Houston, Texas
  - Novartis Investigator Site, Kirkland, Washington
  - Novartis Investigator Site, Seattle, Washington
- Argentina (4):
  - Novartis Investigator Site, Buenos Aires
  - Novartis Investigator Site, Córdoba
  - Novartis Investigator Site, Rosario
  - Novartis Investigator Site, San Miguel de Tucumán
- Canada (5):
  - Novartis Investigator Site, Halifax
  - Novartis Investigator Site, London
  - Novartis Investigator Site, Mississauga
  - Novartis Investigator Site, Montreal
  - Novartis Investigator Site, Ste-Foy
- Czechia (3):
  - Novartis Investigator Site, Brno
  - Novartis Investigative Site, Prague
  - Novartis Investigator Site, Prague
- France (6):
  - Novartis Investigator Site, Brest
  - Novartis Investigator Site, Castelnau-le-Lez
  - Novartis Investigator Site, Chauny
  - Novartis Investigator Site, Paris
  - Novartis Investigator Site, Tarbes
  - Novartis Investigator Site, Vandœuvre-lès-Nancy
- Germany (15):
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Bochum
  - Novartis Investigator Site, Borstel
  - Novartis Investigator Site, Geesthacht
  - Novartis Investigator Site, Hamburg
  - Novartis Investigator Site, Kiel
  - Novartis Investigator Site, Leipzig
  - Novartis Investigator Site, Lübeck
  - Novartis Investigator Site, Mainz
  - Novartis Investigator Site, Marburg
  - Novartis Investigator Site, Neumünster
  - Novartis Investigator Site, Neuss
  - Novartis Investigator Site, Schwetzingen
  - Novartis Investigator Site, Wiesloch
  - Novartis Investigator Site, Wittem
- Hungary (5):
  - Novartis Investigator Site, Debrecen
  - Novartis Investigator Site, Nyíregyháza
  - Novartis Investigator Site, Sopron
  - Novartis Investigator Site, Szombathely
  - Novartis Investigator Site, Tatabánya
- Italy (9):
  - Novartis Investigator Site, Brescia
  - Novartis Investigator Site, Catania
  - Novartis Investigator Site, Modena
  - Novartis Investigator Site, Parma
  - Novartis Investigator Site, Pietra Ligure
  - Novartis Investigator Site, Pisa
  - Novartis Investigator Site, Terni
  - Novartis Investigator Site, Torino
  - Novartis Investigator Site, Trieste
- Novartis Investigator Site, Lima, Peru
- Slovakia (5):
  - Novartis Investigator Site, Bardejov
  - Novartis Investigator Site, Bratislava
  - Novartis Investigator Site, Košice
  - Novartis Investigator Site, Nitra
  - Novartis Investigator Site, Trenčín
- Spain (13):
  - Novartis Investigator Site, Alicante
  - Novartis Investigator Site, Barcelona
  - Novartis Investigator Site, Begonte
  - Novartis Investigator Site, Cadiz
  - Novartis Investigator Site, Cáceres
  - Novartis Investigator Site, Granollers
  - Novartis Investigator Site, Hostalets de Balenyà
  - Novartis Investigator Site, Illescas
  - Novartis Investigative Site, L'Hospitalet de Llobregat
  - Novartis Investigator Site, Mataró
  - Novartis Investigator Site, Oviedo
  - Novartis Investigator Site, Seville
  - Novartis Investigator Site, Valencia
- Turkey (Türkiye) (4):
  - Novartis Investigator Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigator Site, Istanbul
  - Novartis Investigator Site, Izmir

RESULTS

PARTICIPANT FLOW:
Groups:
- Indacaterol 300 μg: Patients received indacaterol 300 μg delivered via a single dose dry powder inhaler (SDDPI) once daily (od) in the morning (between 7:00 and 11:00 AM). In addition to indacaterol 300 μg, patients received indacaterol and salmeterol placebo inhalations in the morning and salmeterol placebo inhalation in the evening (between 7:00 and 11:00 PM). Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Indacaterol 600 μg: Patients received indacaterol 600 μg (2 x 300 μg capsules) delivered via single dose dry powder inhalers (SDDPI) once daily (od) in the morning (between 7:00 and 11:00 AM). In addition to indacaterol 600 μg, patients received salmeterol placebo inhalation in the morning and the evening (between 7:00 and 11:00 PM). Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Salmeterol 50 μg: Patients received salmeterol 50 μg delivered via the salmeterol proprietary dry powder inhalation device bis in die (bid, twice daily), once in the morning (between 7:00 and 11:00 AM) and once in the evening (between 7:00 and 11:00 PM). In addition to salmeterol 50 μg, patients received 2 indacaterol placebo inhalations in the morning. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
Period: Overall Study
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Started | 268 | 268 | 269
Completed | 225 | 225 | 238
Not Completed | 43 | 43 | 31
Not completed — Adverse Event | 12 | 17 | 8
Not completed — Subject withdrew consent | 12 | 9 | 12
Not completed — Protocol deviation | 8 | 12 | 5
Not completed — Lost to Follow-up | 5 | 3 | 1
Not completed — Unsatisfactory therapeutic effect | 2 | 2 | 2
Not completed — Death | 2 | 0 | 0
Not completed — Abnormal test procedure result(s) | 1 | 0 | 0
Not completed — Administrative problems | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg | Total
Number analyzed (Participants) | 268 | 268 | 269 | 805
Age Continuous [Mean (Standard Deviation); unit: years] | 43.5 (15.84) | 44.5 (15.19) | 42.5 (15.24) | 43.5 (15.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 175 | 164 | 490
  Male | 117 | 93 | 105 | 315

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With at Least 1 Adverse Event During the 26 Weeks of the Study
Description: Adverse events include asthma exacerbations. An asthma exacerbation was defined as a worsening of asthma as judged clinically significant by the physician, requiring treatment with rescue oral or intravenous (IV) corticosteroids. Asthma worsening that required treatment with inhaled or nebulized short-acting β2-agonists or an increase in inhaled corticosteroids only was not considered an asthma exacerbation.
Time Frame: Baseline (Day 1) to end of study (Week 26)
Population: Safety population: All patients who received at least one dose of study drug.
Measure: Number; unit: Percentage of patients
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 268 | 268 | 269
Percentage of patients | 54.9 | 66.4 | 67.3

2. Primary Outcome: Systolic Blood Pressure 1 Hour Post-dose at Day 1
Description: Systolic blood pressure measurements (in millimeters of mercury, mmHg) were made 1 hour post-dose after the patient had rested in the sitting position for at least 10 minutes. Measurements were made using an inflatable cuff around the upper arm. The analysis included baseline systolic blood pressure and forced expiratory volume in 1 second (FEV1) pre-dose and 30 minutes post-dose of salbutamol/albuterol during screening as covariates.
Time Frame: Day 1
Population: Safety population: All patients who received at least one dose of study drug. Participants with observations at Day 1 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 263 | 264 | 264
mmHg | 122.79 (0.605) | 122.60 (0.605) | 122.56 (0.606)

3. Primary Outcome: Systolic Blood Pressure 1 Hour Post-dose at Week 12
Description: Systolic blood pressure measurements (in millimeters of mercury, mmHg) were made 1 hour post-dose after the patient had rested in the sitting position for at least 10 minutes. Measurements were made using an inflatable cuff around the upper arm. The analysis included baseline systolic blood pressure and FEV1 pre-dose and 30 minutes post-dose of salbutamol/albuterol during screening as covariates.
Time Frame: Week 12
Population: Safety population: All patients who received at least one dose of study drug. Participants with observations at week 12 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 238 | 237 | 244
mmHg | 120.29 (0.802) | 121.98 (0.809) | 122.02 (0.801)

4. Primary Outcome: Diastolic Blood Pressure 1 Hour Post-dose at Day 1
Description: Diastolic blood pressure measurements (in millimeters of mercury, mmHg) were made 1 hour post-dose after the patient had rested in the sitting position for at least 10 minutes. Measurements were made using an inflatable cuff around the upper arm. Phase V Korotkoff sounds were used for determination of diastolic pressure. The analysis included baseline diastolic blood pressure and FEV1 pre-dose and 30 minutes post-dose of salbutamol/albuterol during screening as covariates.
Time Frame: Day 1
Population: Safety population: All patients who received at least one dose of study drug. Participants with observations at Day 1 were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 263 | 264 | 264
mmHg | 76.67 (0.484) | 76.55 (0.484) | 77.08 (0.485)

5. Primary Outcome: Diastolic Blood Pressure 1 Hour Post-dose at Week 12
Description: as for outcome 4
Time Frame: Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 238 | 237 | 244
mmHg | 75.38 (0.576) | 76.11 (0.580) | 76.96 (0.575)

6. Primary Outcome: Corrected QT (QTc) Interval Using Fridericia's Formula Measured 1 Hour Post-dose at Day 1
Description: The QTc interval (in milliseconds, ms) is calculated from electrocardiogram (ECG) data collected 1 hour post-dose using Fridericia's formula: QTc = QT/RR^0.33. QTc is the interval between the Q and T waves corrected for heart rate and RR is the interval between two R waves. ECGs included all 12 standard leads and a Lead II rhythm strip of at least 10-second duration. All results were sent to a central laboratory for review by a cardiologist. The analysis included baseline QTc interval and FEV1 pre-dose and 30 minutes post-dose of salbutamol/albuterol during screening as covariates.
Time Frame: Day 1
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ms
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 265 | 265 | 265
ms | 404.46 (0.706) | 404.97 (0.704) | 405.05 (0.706)

7. Primary Outcome: Corrected QT (QTc) Interval Using Fridericia's Formula Measured 1 Hour Post-dose at Week 12
Description: as for outcome 6
Time Frame: Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ms
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 238 | 236 | 242
ms | 404.93 (0.970) | 407.78 (0.979) | 406.98 (0.967)

8. Primary Outcome: Corrected QT (QTc) Interval Using Fridericia's Formula Measured 1 Hour Post-dose at Week 21
Description: as for outcome 6
Time Frame: Week 21
Population: Safety population: All patients who received at least one dose of study drug. Participants with observations at week 21 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: ms
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 227 | 228 | 237
ms | 406.41 (1.005) | 407.49 (1.014) | 407.23 (0.995)

9. Primary Outcome: 24 Hour Mean Heart Rate Determined From ECG Holter Monitoring at Week 12
Description: Continuous 24 hour electrocardiography (Holter monitoring) was conducted in a subset of patients at designated study centers, and was used to calculate the mean heart rate (in beats per minute, bpm). Patients returned the Holter monitor recorder to the clinic the morning after the 24 hour recording was complete. The results of Holter monitoring were processed centrally. The analysis included baseline 24 hour mean heart rate and FEV1 pre-dose and 30 minutes post-dose of salbutamol/albuterol during screening as covariates.
Time Frame: Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 74 | 75 | 69
bpm | 81.0 (1.10) | 81.7 (1.11) | 80.4 (1.05)

10. Primary Outcome: 24 Hour Mean Heart Rate Determined From ECG Holter Monitoring at Week 26
Description: as for outcome 9
Time Frame: Week 26
Population: Safety population: All patients who received at least one dose of study drug. Participants with observations at week 26 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 64 | 65 | 63
bpm | 79.4 (0.96) | 81.0 (0.96) | 79.2 (0.96)

11. Primary Outcome: Serum Potassium 1 Hour Post-dose at Day 1
Description: Serum potassium (in millimoles per liter, mmol/L) was measured from venous blood samples. Samples were sent to a central laboratory for analysis. The analysis included baseline serum potassium and FEV1 pre-dose and 30 minutes post-dose of salbutamol/albuterol during screening as covariates.
Time Frame: Day 1
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 266 | 262 | 257
mmol/L | 4.30 (0.022) | 4.24 (0.023) | 4.32 (0.023)

12. Primary Outcome: Serum Potassium 1 Hour Post-dose at Week 12
Description: as for outcome 11
Time Frame: Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 235 | 233 | 241
mmol/L | 4.31 (0.025) | 4.29 (0.025) | 4.33 (0.025)

13. Primary Outcome: Blood Glucose 1 Hour Post-dose at Day 1
Description: Blood glucose (in millimoles per liter, mmol/L) was measured from venous blood samples. Samples were sent to a central laboratory for analysis. The analysis included baseline blood glucose and FEV1 pre-dose and 30 minutes post-dose of salbutamol/albuterol during screening as covariates.
Time Frame: Day 1
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 266 | 265 | 258
mmol/L | 5.24 (0.061) | 5.45 (0.061) | 5.21 (0.062)

14. Primary Outcome: Blood Glucose 1 Hour Post-dose at Week 12
Description: as for outcome 13
Time Frame: Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 235 | 234 | 241
mmol/L | 5.27 (0.068) | 5.38 (0.069) | 5.23 (0.068)

15. Primary Outcome: Percentage of Patients With Clinically Significant Asthma Exacerbations During the 26 Weeks of the Study
Description: A clinically significant asthma exacerbation was defined as a worsening of asthma as judged clinically significant by the physician, requiring treatment with systemic corticosteroids. This includes events recorded on the asthma exacerbation clinical report form (CRF) page and events recorded on the adverse events CRF page with "asthma" as a key word in the preferred term.
Time Frame: Baseline (Day 1) to end of study (Week 26)
Population: Intent-to-treat (ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of patients
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 268 | 268 | 269
Percentage of patients
  0 exacerbations | 92.9 | 89.9 | 90.0
  1 exacerbation | 5.6 | 9.3 | 8.6
  2 exacerbations | 0.7 | 0.7 | 1.5
  3 exacerbations | 0.7 | 0.0 | 0.0

16. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose at Week 12 + 1 Day, Day 85
Description: FEV1 (in liters, L) was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose at Week 12, Day 85. The analysis included baseline FEV1 and FEV1 pre-dose and 30 minutes post-dose of salbutamol during screening as covariates.
Time Frame: 24 hours post-dose at Week 12 + 1 day, Day 85
Population: Intent-to-treat (ITT) population: All randomized patients who received at least 1 dose of study drug. Participants with observations at Day 85 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 258 | 255 | 262
Liters | 2.61 (0.023) | 2.62 (0.023) | 2.54 (0.023)

17. Secondary Outcome: Number of Asthma Exacerbations Per Patient (Without Imputation) During the 26 Weeks of the Study
Description: An asthma exacerbation was defined as a worsening of asthma as judged clinically significant by the physician, requiring treatment with rescue oral or intravenous (IV) corticosteroids. The number of asthma exacerbations includes events recorded on the asthma exacerbation clinical report form (CRF) page and events recorded on the adverse events CRF page with "asthma" as a key word in the preferred term.
Time Frame: Baseline (Day 1) to end of study (Week 26)
Population: Intent-to-treat (ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Asthma exacerbations
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Number analyzed (Participants) | 268 | 268 | 269
Asthma exacerbations | 0.17 (0.561) | 0.19 (0.512) | 0.19 (0.494)

ADVERSE EVENTS:
Time Frame: Baseline to the end of the study (Week 26)
Description: Safety population: All patients who received at least one dose of study drug.
Arm/Group | Indacaterol 300 μg | Indacaterol 600 μg | Salmeterol 50 μg
Serious Adverse Events (participants affected / at risk) | 5/268 | 11/268 | 8/269
Other Adverse Events (participants affected / at risk) | 86/268 | 105/268 | 101/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 300 μg (N=268) | Indacaterol 600 μg (N=268) | Salmeterol 50 μg (N=269)
Splenic cyst (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Sudden death (General disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 1
Stress (Psychiatric disorders) | 1 | 0 | 0
Analgesic asthma syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 300 μg (N=268) | Indacaterol 600 μg (N=268) | Salmeterol 50 μg (N=269)
Bronchitis (Infections and infestations) | 10 | 13 | 16
Nasopharyngitis (Infections and infestations) | 20 | 22 | 26
Upper respiratory tract infection (Infections and infestations) | 17 | 27 | 18
Headache (Nervous system disorders) | 14 | 18 | 20
Asthma (Respiratory, thoracic and mediastinal disorders) | 30 | 39 | 40
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 29 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.